CLINICAL TRIAL: NCT04629976
Title: Randomized, Open-Label, Active Comparator, Multiple Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-Hepatitis B Virus (HBV) Activity of NCO-48 Fumarate in Treatment-Naive Adults With Chronic HBV Infection
Brief Title: Activity of NCO-48 Fumarate in Treatment-Naive Adults With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nucorion Pharmaceuticals, Inc. (Industry)
Collaborators: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCO48F-02
Record Dates: First submitted 2020-11-04; First posted 2020-11-16 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: After Screening procedures, eligible subjects will be randomized 1:1:1 to receive either open-label NCO-48 Fumarate 4 mg (2 x 2 mg) or 20 mg (2 x 10 mg), or open-label TAF 25 mg for 28 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NCO-48 Fumarate 4 mg (Experimental): Eligible subjects will be randomized 1:1:1 to receive either open-label NCO-48 Fumarate 4 mg or 20 mg, or open-label TAF 25 mg for 28 days.
  Interventions: Drug: NCO-48 Fumarate 4 mg
- NCO-48 Fumarate 20 mg (Experimental): Eligible subjects will be randomized 1:1:1 to receive either open-label NCO-48 Fumarate 4 mg or 20 mg, or open-label TAF 25 mg for 28 days.
  Interventions: Drug: NCO-48 Fumarate 20 mg
- Tenofovir alafenamide 25 mg (Active Comparator): Eligible subjects will be randomized 1:1:1 to receive either open-label NCO-48 Fumarate 4 mg or 20 mg, or open-label TAF 25 mg for 28 days.
  Interventions: Drug: Tenofovir Alafenamide 25 mg

INTERVENTIONS:
Drug: NCO-48 Fumarate 4 mg — 2 x 2mg NCO-48 Fumarate over 28 days of therapy
  Arms: NCO-48 Fumarate 4 mg
Drug: NCO-48 Fumarate 20 mg — 2 x 10 mg NCO-48 Fumarate over 28 days of therapy
  Arms: NCO-48 Fumarate 20 mg
Drug: Tenofovir Alafenamide 25 mg — 25 mg over 28 days of therapy
  Other Names: Vemlidy ®
  Arms: Tenofovir alafenamide 25 mg

SUMMARY:
This is an open-label study evaluating multiple doses of NCO-48 Fumarate versus tenofovir alafenamide (TAF).

DETAILED DESCRIPTION:
This is a randomized, open-label, active comparator, multiple oral dose study to evaluate the safety, tolerability, pharmacokinetics, and anti-hepatitis B virus (HBV) activity of NCO-48 Fumarate in treatment-naive adults with chronic HBV infection. This study will evaluate the safety, viral kinetics, and antiviral activity of 2 different doses of NCO-48 Fumarate over 28 days of therapy. In addition, the study will evaluate the antiviral activity of an optimal dose of NCO-48 Fumarate versus 25 mg tenofovir alafenamide (TAF) over 28 days of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects between 18 and 65 years of age
* Female subjects of non-childbearing potential must be surgically sterile or postmenopausal at the Screening Visit
* Female subjects of childbearing potential who are sexually active with a non-sterile male partner must be using a medically acceptable form of birth control for the duration of the study and for 30 days after the last dose of study drug and must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test upon admission to the study site
* HBV treatment-naive or treatment-experienced with (pegylated or non pegylated) interferon alpha (must have ended at least 6 months prior to the Screening Visit)
* Screening plasma HBV DNA ≥ 2x10^3 IU/mL
* Positive for serum hepatitis B surface antigen for more than 6 months
* Estimated creatinine clearance (CLCr) ≥ 70 mL/min
* Serum transaminase activity (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] levels) <10 x the upper limit of normal
* Compensated liver disease with normal prothrombin time/international normalized ratio, hematology, albumin, bilirubin (unless subject has Gilbert's disease). Serum AST and/or ALT levels may be normal or elevated
* Body mass index within the range of 18.5 to 35 kg/m2, inclusive, and body weight >45 kg
* Normal vital signs, without any clinically significant abnormalities at the Screening Visit
* Subjects who have normal or abnormal clinically insignificant clinical laboratory assessments as considered by the Investigator from pre-treatment blood tests to assess hematology, liver (except for serum AST and/or ALT levels) and renal biochemistry, urinalysis, and drug screen
* Normal 12-lead electrocardiogram (ECG), with no clinically significant abnormalities of rate, rhythm, or conduction and including normal heart rate-corrected QT interval segment time at the Screening Visit

Exclusion Criteria:

* Received treatment with TFV disoproxil fumarate or TAF (including clinical study experience)
* Positive for hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* History or presence of asthma or other pulmonary disease, thyroid disease, or other liver disease
* Hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism, or excretion of study drug, or would place the subject at increased risk
* Abnormal laboratory values that are considered clinically significant
* Have used medication, other than topical products without significant systemic absorption, hormonal contraceptives, or hormone replacement therapy and thyroid medication for at least 6 months
* Unwilling to refrain from consumption of alcohol within 48 hours prior to each dose of study drug and during the inpatient period, or have a history of significant alcohol abuse within 1 year prior to Screening
* Positive urine drug screen, or positive alcohol breath test at Screening or upon admission to the study site
* Use of illicit drugs within 3 months prior to the Screening Visit or hard drugs within 1 year prior to the Screening Visit, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction
* Women who are breastfeeding or have a positive pregnancy test at the Screening Visit or at any time during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Change in hepatitis B virus (HBV) DNA | Up to Week 4
  Time-weighted average change from baseline through Week 4 in plasma HBV DNA (log10 IU/mL) for NCO-48 Fumarate 4 and 20-mg.

SECONDARY OUTCOMES:
Change in HBV DNA for tenofovir alafenamide (TAF) | Up to Week 4
  Comparing the short-term antiviral activity of NCO-48 Fumarate with TAF 25 mg. This is measured by time-weighted average change from baseline through Week 4 in plasma HBV DNA (log10 IU/mL) for TAF.
Incidence of Treatment-Emergent Adverse Events | Up to week 4
  Safety and tolerability is measured by the incidence of treatment-emergent adverse events.
NCO-48 Fumarate Area Under the Concentration -Time Curve (AUC) | Up to week 4
  Blood samples are to be collected at designated time points for the determination of the NCO-48 Fumarate AUC.
NCO-48 Fumarate Maximum Plasma Concentration (Cmax) | Up to week 4
  Blood samples are to be collected at designated time points for the determination of the NCO-48 Fumarate Cmax.
Tenofovir (TFV) Area under the Concentration-Time Curve (AUC) | Up to week 4
  Blood samples are to be collected at designated time points for the determination of TFV AUC.
TFV Maximum Plasma Concentration (Cmax) | Up to week 4
  Blood samples are to be collected at designated time points for the determination of TFV Cmax.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Marschke, Study Director — Ligand Pharmaceuticals
Locations (1):
- National Institute of Clinical Research, Inc, Monterey Park, California, United States